CLINICAL TRIAL: NCT04114214
Title: Development of an Objective Sepsis Identification Tool to Study Sepsis Epidemiology: a Single Center Retrospective Cohort Study
Brief Title: Objective Sepsis Identification Tool to Study Sepsis Epidemiology
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lowell Ling, Clinical Lecturer, Chinese University of Hong Kong
Other Study IDs: 2019.214
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with suspected infection or sepsis: All patients admitted with suspected infection or sepsis from January 2018 to February 2018 at Prince of Wales Hospital

SUMMARY:
Globally, sepsis affects an estimated 31.5 million people and accounts for 5.3 million deaths each year. This calculation is based on data from western high income countries only. The purpose of this study is to develop an objective sepsis identification tool using electronic health records to study the epidemiology of sepsis in Hong Kong.

DETAILED DESCRIPTION:
Globally, sepsis affects an estimated 31.5 million people and accounts for 5.3 million deaths each year. The incidence of sepsis is increasing and is now a more common cause for hospital admission than acute myocardial infarction and stroke.

However this apparent improvement in sepsis outcomes may also be due to changes in definition and reporting of sepsis. The latest Sepsis-3 definition outlines sepsis as life-threatening organ dysfunction due to dysregulated host response to infection. Trends on sepsis incidence and outcome were based on previous definitions of sepsis. Furthermore, changes in coding practices and documentation for hospital claims may cause misleading changes in incidence and outcomes. Electronic health record clinical data provides more reliable data on sepsis epidemiology than diagnostic coding accounts for. Our understanding of sepsis epidemiology is based on studies from high income western countries. Even within these countries, health expenditure and resources vary which may affect sepsis outcomes. Current data on the burden of sepsis from the rest of the world is insufficient. Hong Kong is well poised to provide these lacking data on the epidemiology of sepsis. More than 90% of inpatient care is provided by the public healthcare system and would be captured by the electronic Clinical Management System. The purpose of this study is to develop an objective sepsis identification tool using electronic health records to study the epidemiology of sepsis in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* January 2018 to February 2018 adult inpatients at Prince of Wales Hospital
* 1st microbiological culture tests during hospital admission

Exclusion Criteria:

* duplicated microbiological sampling
* missing values for sequential organ failure assessment score calculation
* microbiological tests were for screening only (methicillin-resistant staphylococcus aureus swabs, vancomycin resistant Enterococci rectal swab)
* antibiotics not started 2 days before or after first microbiological sampling
* antibiotics duration less than 4 days unless death
* not given antibiotics on discharge if given less than 4 days antibiotics in hospital

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to Prince of Wales Hospital in Hong Kong between January 2018 to February 2018 with suspected infection.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Classification of Sepsis | within 2 days of microbiological sampling
  comparison with clinician review of case notes

SECONDARY OUTCOMES:
Organ Dysfunction | within 2 days of microbiological sampling
  Estimated Organ Dysfunction from sequential organ failure assessment
28 Day Mortality | 28 days
  28 Day Mortality of Hospital Episode
Hospital Length of Stay | 1 year
  Hospital Length of Stay of Hospital Episode

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu YZ, Chu R, Lee A, Gomersall CD, Zhang L, Gin T, Chan MTV, Wu WKK, Ling L. A surveillance method to identify patients with sepsis from electronic health records in Hong Kong: a single centre retrospective study. BMC Infect Dis. 2020 Sep 7;20(1):652. doi: 10.1186/s12879-020-05330-x. PMID 32894059